CLINICAL TRIAL: NCT06139211
Title: A Phase Ib/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of JS015 Combination Therapy in Patients With Advanced Solid Tumors
Brief Title: A Phase Ib/II Study Of JS015 Combination Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS015-002-Ib/II-GI
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab; Paclitaxel; Irinotecan; Capecitabine; Oxaliplatin; Bevacizumab; Fluorouracil; Leucovorin; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1: esophogeal squamous carcinoma (Experimental): In Cohort 1, patients will be treated with JS015 in combination with paclitaxel or irinotecan
  Interventions: Biological: JS015; Biological: Paclitaxel; Drug: Irinotecan
- Cohort 2: gastric cancer (Experimental): In Cohort 2, patients will be treated with JS015 in combination with paclitaxel
  Interventions: Biological: JS015; Biological: Paclitaxel
- Cohort 3: gastric cancer (Experimental): In Cohort 3, patients will be treated with JS015 in combination with toripalimab and XELOX
  Interventions: Biological: JS015; Biological: Toripalimab; Drug: Capecitabine; Drug: Oxaliplatin
- Cohort 4: colorectal cancer (Experimental): In Cohort 4, patients will be treated with JS015 plus bevacizumab in combination with XELOX or FOLFIRI
  Interventions: Biological: JS015; Drug: Irinotecan; Drug: Capecitabine; Drug: Oxaliplatin; Biological: Bevacizumab; Drug: Fluorouracil; Drug: Leucovorin
- Cohort 5: pancreatic cancer (Experimental): In Cohort 5, patients will be treated with JS015 in combination with toripalimab, albumin-bound paclitaxel and gemcitabine
  Interventions: Biological: JS015; Biological: Toripalimab; Drug: Gemcitabine; Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Biological: JS015 — JS015 will be administered intravenously (IV) on days 1 and 15 every 28 day cycle, or day 1 every 21 day cycle, based on different combined chemotherapy.
Biological: Toripalimab — Toripalimab will be administered intravenously (IV) on day 1 every 21 day cycle.
  Arms: Cohort 3: gastric cancer; Cohort 5: pancreatic cancer
Biological: Paclitaxel — Paclitaxel will be administered intravenously (IV) on day 1 every 21 day cycle.
  Arms: Cohort 1: esophogeal squamous carcinoma; Cohort 2: gastric cancer
Drug: Irinotecan — Irinotecan will be administered intravenously (IV) on days 1 and 15 every 28 day cycle.
  Arms: Cohort 1: esophogeal squamous carcinoma; Cohort 4: colorectal cancer
Drug: Capecitabine — Capecitabin will be administered orally twice daily from day 1 to 14 every 21 day cycle.
  Arms: Cohort 3: gastric cancer; Cohort 4: colorectal cancer
Drug: Oxaliplatin — Oxaliplatin will be administered intravenously (IV) on day 1 every 21 day cycle.
  Arms: Cohort 3: gastric cancer; Cohort 4: colorectal cancer
Biological: Bevacizumab — Bevacizumab of 5mg/kg will be administered intravenously (IV) on days 1 and 15 every 28 day cycle, or7.5mg/kg on day 1 every 21 day cycle, based on different combined chemotherapy.
  Arms: Cohort 4: colorectal cancer
Drug: Fluorouracil — Fluorouracil will be administered intravenously (IV) on days 1 and 15 every 28 day cycle.
  Arms: Cohort 4: colorectal cancer
Drug: Leucovorin — Leucovorin will be administered intravenously (IV) on days 1 and 15 every 28 day cycle.
  Arms: Cohort 4: colorectal cancer
Drug: Gemcitabine — Gemcitabine will be administered intravenously (IV) on days 1 and 8 every 21 day cycle.
  Arms: Cohort 5: pancreatic cancer
Drug: Albumin-Bound Paclitaxel — Albumin-bound paclitaxel will be administered intravenously (IV) on days 1 and 8 every 21 day cycle.
  Arms: Cohort 5: pancreatic cancer

SUMMARY:
This is a phase Ib/II, open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of JS015 combination therapy in patients with advanced solid tumors. The Recommended dose for phase II trial （RP2D） will be determined based on the safety, tolerability, pharmacokinetics and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the following criteria for each indication cohort:

1. Esophageal cancer cohort, patients with histologically or cytologically confirmed esophageal squamous cell carcinoma with locally advanced unresectable or with distant metastasis, who progressed during or after prior first-line PD-(L)1 antibody and platinum-based chemotherapy;
2. Gastric cancer cohort, patients with histologically or cytologically confirmed gastric/gastroesophageal junction adenocarcinoma with locally advanced unresectable or distant metastases, HER2-negative, who progressed during or after prior first-line PD-(L)1 antibody and platinum-based chemotherapy;
3. 1L gastric cancer cohort, patients with histologically or cytologically confirmed gastric/gastroesophageal junction adenocarcinoma with HER2-negative results and no prior systemic antitumor therapy;
4. Colorectal cancer cohort, patients with histologically confirmed adenocarcinoma of the colon or rectum, who progressed during or after first-line 5-FU-based combination therapy;
5. Pancreatic cancer cohort, patients with histologically or cytologically confirmed locally advanced unresectable or distant metastatic pancreatic ductal adenocarcinoma, who have not received any previous systemic antitumor therapy 2 . Eastern Cooperative Oncology Group (ECOG) 0 or 1; 3. Life expectancy >=12 weeks; 4. At least one measurable lesion according to RECIST 1.1; 5. Adequate organ function;

Exclusion Criteria:

1. Leptomeningeal metastases and /or active brain metastases;
2. Pleural, peritoneal, or pericardial effusion with clinical symptoms or requiring repeated management (puncture, drainage, etc.);
3. History of interstitial lung disease or a previous history of noninfectious pneumonia with corticosteroid therapy, or evidence of active pneumonia on screening imaging;
4. History of immunodeficiency;
5. History of serious cardiovascular and/or cerebrovascular diseases;
6. History of abdominal or tracheo-esophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months before the first dose of administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
incidence of dose-limiting toxicity （DLT） | 2 Years
  incidence and severity of DLT
incidence of adverse event（AE） | 2 Years
  adverse events (AE)
Recommended dose for phase II trial RP2D | 2 Years
  Recommended dose for phase II trial

SECONDARY OUTCOMES:
Peak concentration (Cmax) | 2 years
  The highest plasma drug concentration that can be achieved after medication
time to peak concentration（Tmax） | 2 years
  The time it takes for the drug to reach its maximum concentration (Cmax) in the plasma after administration
elimination half life（t1/2） | 2 years
  The time it takes for the concentration of the drug in the plasma to be reduced by 50%
immunogenicity | 2 years
  Incidence of Anti-Drug Antibody (ADA)
Objective response rate (ORR) based on Response Evaluation Criteria In Solid Tumors 1.1 (RECIST1.1) | 2 years
  Defined as the proportion of subjects who achieved partial response (PR) or complete response (CR)
Progression free survival (PFS) | 2 years
  The time from first dose to Disease progression or death
overall survival (OS) | 2 years
  The time from first dose to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No